CLINICAL TRIAL: NCT00247026
Title: A Pilot Study to Determine the Clinical Efficacy of Coenzyme Q10 And Curcumin in Patients With Myelodysplastic Syndromes
Brief Title: The Efficacy of Coenzyme Q10 And Curcumin in Patients With Myelodysplastic Syndromes
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 385-mds 1-HMO-CTIL; mds 1
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplasia; curcumin; coenzyme Q10; cytopenia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Cytopenia | interventions — Curcumin; coenzyme Q10

INTERVENTIONS:
Drug: curcumin; coenzyme q10

SUMMARY:
To determine the clinical effects of coenzyme Q10 and Curcumin in improving the cytopenias of patients with myelodysplastic syndromes. we propose to explore the efficacy of the natural compounds curcumin and CoQ10 in MDS because these two agents possess many of the effects that are desirable in MDS.

ELIGIBILITY:
Inclusion Criteria:

* MDS patients with RA, RARS or RAEB will be eligible for treatment with CoQ10 as long as their IPSS score ≤ 1.5.

Exclusion Criteria:

* Pregnant women and nursing women will be excluded.
* History of clinically significant liver or kidney disease.
* ECOG>2
* IPSS score >1.5
* Poorly controlled diabetes mellitus, hypertension, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to the protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2007-04

PRIMARY OUTCOMES:
major hematologic improvement in any lineage

SECONDARY OUTCOMES:
Time to disease progression
Overall and progression-free survival
Cytogenetic response

CONTACTS AND LOCATIONS:
Overall Officials: moshe e gatt, dr, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel